CLINICAL TRIAL: NCT02736045
Title: The Impact of Work Burnout on Sleep Quality and Negative Emotions in Medical Residents: An Intervention for Improving Wellbeing in Graduate Medical Education
Brief Title: Ameliorating Work Burnout and Medical Residents
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Period Ended / Not Completed
Sponsor: Larkin Community Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: LCH-1-032015
Record Dates: First submitted 2015-04-27; First posted 2016-04-13 (Estimated); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Burnout, Professional; Depression; Stress; Anxiety; Distress
MeSH Terms: conditions — Burnout, Professional; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Sham control. Subjects will be asked to write a journal (per week).
- emWave (Experimental): Our approach will be to test the impact of a behavioral intervention through a smartphone application, emWave software, which will be provided to all our subjects. The intervention (emWave) is a tool that reduces stress by allowing individuals to be less reactive, think clearly, and make good decisions, especially under pressure. Fifty medical residents with high burnout symptoms will be randomized to receive an 8-week intervention.
  Interventions: Device: emWave

INTERVENTIONS:
Device: emWave — Our approach will be to test the impact of this intervention through a smartphone application, emWave software, which will be provided to all our subjects. emWave is a tool that reduces stress by allowing individuals to be less reactive, think clearly, and make good decisions, especially under pressure. Fifty medical residents with high burnout symptoms will be randomized to receive an 8-week intervention (emWave - computer based resilience training program).
  Other Names: INT
  Arms: emWave

SUMMARY:
Prior research has demonstrated that during residency years, in particular training to obtain a medical specialty, work burnout is a very prevalent problem. Work burnout is defined as a syndrome of dysfunction in three domains, emotional exhaustion, depersonalization, and a reduced sense of personal accomplishment. (Maslach et. al., 1981). Often, burnout has been associated with poor sleep quality and negative affectivity, such as depression and anxiety. In fact, our preliminary data demonstrate that burnout in medical residents affects sleep quality, and increases negative emotions. Strikingly, burnout in medical residents negatively impacts working performance as well as patient-physician interactions, and hence may affect the quality of health care. However, lacking are studies aimed at understating how work burnout affects cognitive performance and decision making in medical residents. The proposed study will provide essential groundwork in demonstrating the link between burnout and impaired cognitive performance. In addition, the proposed study will demonstrate feasibility for a future trial to test whether an intervention, emWave, integrating a computer based stress management (resilience training), can have a positive impact on residents with high burnout symptoms. The amelioration of psychological risk factors in medical residents may lead to improved physician-patient relationships in the service of improved quality of care.

DETAILED DESCRIPTION:
Background: Burnout during residency years, in particular training to obtain a medical specialty, has been well recognized. Often, burnout has been associated with poor sleep quality and negative affectivity, such as depression. However, aspects of positive emotion that have been linked to improved physical and mental health, such as trait forgiveness (TF), have been poorly explored.

For instance, according to statistics, depression in residents is as high as twenty-five percent, while residents' suffering from depression with resident burnout (defined as an occupational related syndrome of emotional exhaustion and low sense of professional accomplishment) is as high as seventy-six percent. In fact, first-year residents, with a sense of high well-being, experience great level of burnout and depression by the end of their first year. ( www.aafp.org, Yi M.S. et al. , 2007 ; Shanafelt T.D. et al. ,2002 ; Richman J.A. et. al. , 1992)

There are two specific aims my collaborators and I are focusing on in in this two-phase study:

Specific Aim 1: To explore the impact of work burnout on cognitive performance and psychological functioning in medical residents. Mounting evidence points towards the conclusion that work burnout can have a negative effect on psychological functioning in medical residents. We will test the working hypothesis that work burnout will be associated with poor cognitive performance, poor sleep quality, and high negative affectivity. Our approach is to use self-reported cognitive impairment and cognitive performance tasks designed to measure three basic processes underlying executive control: (i) updating, (ii) inhibition, and (iii) switching. Negative affective symptoms will be measured using validated psychometric scales for depression (Beck Depressive Inventory; BDI), anxiety (State-Trait Anxiety Inventory; STAI), and anger (State-Trait Anger Expression Inventory-2; STAEI-2). Sleep quality will be assessed via the Pittsburgh Sleep Quality Index (PSQI).

Specific Aim 2 - To examine the impact of an 8-week computer based resilience training intervention on work burnout, cognitive performance, and affectivity in medical residents. Our approach will be to test the impact of this intervention through a SmartPhone (e.g Android Phone or Iphone) application, emWave software, which will be provided to all our subjects. emWave is a tool that reduces stress by allowing individuals to be less reactive, think clearly, and make good decisions, especially under pressure. Fifty medical residents with high burnout symptoms will be randomized to receive an 8-week intervention (INT; n=25) or sham control (CON; n=25).

ELIGIBILITY:
Inclusion Criteria:

* Must be a medical resident attending a valid residency program from either Family Medicine, Internal Medicine, Surgery or Psychiatry at Larkin Community Hospital

Exclusion Criteria:

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07-01 (Estimated); Primary Completion 2016-07-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Work Burnout Symptoms ( measured by Maslach Burnout Inventory) (Of note, changes in Work Burnout Symptoms & Findings by Medical Residents will be attempted to be observed) | Change from baseline work burnout symptoms after 8 weeks
  Work Burnout will be measured using the Maslach Burnout Inventory (MBI:Maslach et. al., 1981). The MBI consists of 22 items that are broken up into three dimensions of burnout: a) nine items relating to emotional exhaustion, b) five to depersonalization, and c) eight to personal accomplishment.

SECONDARY OUTCOMES:
Change in Depression ( measured by Epidemiologic Studies Depression Scale) (Of note, changes in Depressive Symptoms by Medical Residents will be attempted to be observed) | Change from baseline depressive-like symptoms after 8 weeks
  Depression will be measured using the 10-item Center for Epidemiologic Studies Depression Scale (CES-D; Radloff 1977, Santor and Coyne 1997).

OTHER OUTCOMES:
Change in Anxiety State ( measured by State-Trait Anxiety Inventory) ( Of note, changes in Anxiety State by Medical Residents will be attempted to be observed) | Change from baseline anxiety state after 8 weeks
  Anxiety will be measured using the 20-item State-Trait Anxiety Inventory (STAI; Spielberger C.D., 2010). Satisfactory reliability (α > .7) has been established in previous research.
Change in Sleep Quality ( measured by Pittsburgh Sleep Quality Index) ( Of note, changes in Sleep Quality by Medical Residents will be attempted to be observed) | Change from baseline sleep quality index after 8 weeks
  Sleep Quality will be measured using the Pittsburgh Sleep Quality Index (PSQI). This instrument is a well-regarded measure in the sleep research literature. It is 19-item measure assessing sleep quality and disturbance over the past month.

CONTACTS AND LOCATIONS:
Overall Officials: John S Samaan, MD MPH, Principal Investigator — Larkin Community Hospital; Marcos Sanchez-Gonzalez, MD PhD, Study Chair — Larkin Community Hospital; Juan D Oms, MD, Study Director — Larkin Community Hospital
Locations (1):
- Larkin Community Hospital, South Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Santor DA, Coyne JC. Shortening the CES-D to improve its ability to detect cases of depression 9(3) : 233-243, 1997.
- [Background] Maslach C, Jackson S. The measurement of experienced burnout. Journal of Organizational Behavior 2(2) 99-113, 1981.
- [Background] Radloff L. The CES-D Scale : A Self-Report Depression Scale for Research in the General Population. Applied Psychological Measurement. 1(3) : 385-401, 1977.
- [Background] Spielberger, CD. State-Trait Anxiety Inventory. Corsini Encyclopedia of Psychology 1, 2010.
- [Background] Yi MS, Mrus JM, Mueller CV, Luckhaupt SE, Peterman AH, Puchalski CM, Tsevat J. Self-rated health of primary care house officers and its relationship to psychological and spiritual well-being. BMC Med Educ. 2007 May 2;7:9. doi: 10.1186/1472-6920-7-9. PMID 17474998
- [Background] Shanafelt TD, Bradley KA, Wipf JE, Back AL. Burnout and self-reported patient care in an internal medicine residency program. Ann Intern Med. 2002 Mar 5;136(5):358-67. doi: 10.7326/0003-4819-136-5-200203050-00008. PMID 11874308
- [Background] Richman JA, Flaherty JA, Rospenda KM, Christensen ML. Mental health consequences and correlates of reported medical student abuse. JAMA. 1992 Feb 5;267(5):692-4. PMID 1731137